CLINICAL TRIAL: NCT04485156
Title: Treatment Shortening of Drug-Sensitive Pulmonary Tuberculosis Using High Dose Rifampicin to 3 Months After Culture Conversion (Hi-DoRi-3): A Phase 3, Multicenter, Randomized, Open-label, Clinical Trial
Brief Title: Treatment Shortening of Drug-Sensitive Pulmonary Tuberculosis Using High Dose Rifampicin (Hi-DoRi-3)
Acronym: Hi-DoRi-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chonnam National University Hospital (Other); National Medical Center, Seoul (Other); Pusan National University Hospital (Other); Pusan National University Yangsan Hospital (Other); Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Severance Hospital (Other); Korean Institute of Tuberculosis (Other); International Tuberculosis Research Center (Other); Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hi-DoRi-3
Record Dates: First submitted 2020-07-06; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; Rifampicin; Treatment; Shortening
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Rifampin; Isoniazid; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Conventional treatment group) (Active Comparator): Will be treated as recommended by Korean Guidelines For Tuberculosis as well as WHO guidelines (e.g. isoniazid, rifampicin, ethambutol, and pyrazinamide for 2 months followed by isoniazid, rifampicin, (and ethambutol)) Duration of the treatment
  - 6 months in total
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Rifampicin
- Arm 2 (High-dose rifampicin group) (Experimental): High-dose rifampicin, isoniazid, and pyrazinamide
  * Rifampicin: 30mg/kg
  * Isoniazid: 300mg/day
  * Pyrazinamide: 1000mg/day (<50kg), 1500mg/day (50-70kg), 2000mg /day (>70kg), till culture conversion Duration of the treatment
  * Till 12 weeks after culture conversion on liquid media
  Interventions: Drug: High-dose rifampicin; Drug: Isoniazid; Drug: Pyrazinamide

INTERVENTIONS:
Drug: High-dose rifampicin — 30mg/kg
  Arms: Arm 2 (High-dose rifampicin group)
Drug: Isoniazid — 300mg
Drug: Pyrazinamide — 20-30mg/kg
Drug: Ethambutol — 15-20mg/kg
  Arms: Arm 1 (Conventional treatment group)
Drug: Rifampicin — 10mg/kg
  Arms: Arm 1 (Conventional treatment group)

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of the regimen including high dose rifampicin for individualized duration (3 months after Culture Conversion) for the treatment of drug-sensitive pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Documented positivity by sputum Xpert MTB/RIF assay
* Administration of current tuberculosis therapy (if any) for no more than 7 days (≤7) at the time of enrolment.

Exclusion Criteria:

* Negative on Xpert MTB/RIF assay
* Resistance to rifampicin as detected by an Xpert MTB/RIF assay
* Known resistance to isoniazid, rifampicin, or pyrazinamide
* HIV positive
* Cancer patient on anti-cancer chemotherapy
* Uncontrolled DM
* Chronic hepatitis, liver cirrhosis
* Any contraindications of drugs to be used

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of unfavorable treatment outcomes between two arms | Within 18 months of randomization

SECONDARY OUTCOMES:
Time to unfavorable treatment outcomes | Within 18 months of randomization
Time to culture conversion on liquid media | Censored at 2 months of treatment
Proportion of participants with treatment success | At the end of treatment
Proportion of participants with relapse of same strain | At the end of study
Time to relapse with same strain | through study completion, 18months after randomization
Occurrence of AEs grade 3 and above | through study completion, 18months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwak N, Kim JY, Kim HJ, Kwon BS, Lee JH, Mok J, Kwon YS, Kang YA, Park Y, Lee JY, Jeon D, Lee JK, Yang JS, Whang J, Kim KJ, Kim YR, Cheon M, Park J, Hahn S, Yim JJ. High-Dose Rifampicin for 3 Months after Culture Conversion for Drug-Susceptible Pulmonary Tuberculosis. Tuberc Respir Dis (Seoul). 2025 Jan;88(1):170-180. doi: 10.4046/trd.2024.0099. Epub 2024 Sep 27. PMID 39343425
- [Derived] Kwak N, Jeon D, Park Y, Kang YA, Kim KJ, Kim YR, Kwon BS, Kwon YS, Kim HJ, Lee JH, Lee JY, Lee JK, Mok J, Cheon M, Park J, Hahn S, Yim JJ. Treatment shortening of drug-sensitive pulmonary tuberculosis using high-dose rifampicin for 3 months after culture conversion (Hi-DoRi-3): a study protocol for an open-label randomized clinical trial. Trials. 2022 Aug 17;23(1):666. doi: 10.1186/s13063-022-06631-z. PMID 35978342